CLINICAL TRIAL: NCT02393417
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Varying Regimens of CANDIN for Treatment of Common Warts (Verruca Vulgaris)
Brief Title: Safety and Efficacy of Varying Regimens of CANDIN for Treatment of Common Warts (Verruca Vulgaris)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nielsen BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CFW-2D
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Warts
Keywords: Verruca vulgaris; Common Warts
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 0.3 mL of CANDIN administered intralesionally in the largest common wart
  Interventions: Biological: CANDIN
- Cohort 2 (Experimental): 0.5 mL of CANDIN administered intralesionally in the largest common wart
  Interventions: Biological: CANDIN
- Cohort 3 (Experimental): 0.3 mL of CANDIN administered intralesionally in up to 4 warts at the same visit (up to 1.2 mL total injected volume)
  Interventions: Biological: CANDIN
- Pooled Placebo (Placebo Comparator): 0.3 mL or 0.5 mL administered intralesionally in the largest common wart, or 0.3 mL administered intralesionally in up to 4 warts at the same visit (up to 1.2 mL total injected volume)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CANDIN — Candida albicans Skin Test Antigen for Cellular Hypersensitivity
  Arms: Cohort 1; Cohort 2; Cohort 3
Other: Placebo — 0.9% Sodium Chloride Injection USP (non-preserved)
  Arms: Pooled Placebo

SUMMARY:
This is a placebo-controlled, double-blind (subject, Investigator, and site staff with the exception of unblinded dedicated staff to handle study medication), phase 2a study with 3 dose cohorts, randomized (concealed) to CANDIN or placebo (3:1). Main study will be up to 20 weeks (10 doses administered every other week) or until a subject has complete resolution of all injectable common warts. Subjects who cannot tolerate dosing every 2 weeks due to a local tolerance issue may be injected at 3-week intervals for up to 10 doses, increasing the length of the study to 29 weeks. Subjects will be followed for 4 months after final injection(s) for evidence of new or reoccurring warts and for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between the ages of 18 and 65 years inclusively at time of consent
2. Subjects presenting with 3 to 20 injectable common warts (verruca vulgaris) for at least 12 weeks at the time of the Baseline Visit
3. Subject's common warts for injection must measure between 3 and 20 mm at Baseline Visit and be located on hands, feet (excluding soles), limbs, and/or trunk. Flat, plantar, facial, periungual, genital warts or warts in region of pre-existing inflammatory condition are excluded from injection
4. Subjects enrolled into Cohort 3 must have common warts for injection in at least 2 different anatomical regions defined as: left arm, right arm, left hand, right hand, left leg, right leg, left foot (excluding sole), right foot (excluding sole) and torso
5. Subject, male or female is willing to use effective contraceptive method for at least 30 days before the Baseline Visit and at least 30 days after the last study drug administration unless not of childbearing potential as defined as post-menopausal for at least 2 years (females) or surgically sterile (tubal ligation, oophorectomy, or hysterectomy for females, and vasectomy for males). The only contraceptive use exceptions would be individuals in exclusive same sex partnerships and individuals who agree to remain non-sexually active for the duration of the study. Acceptable contraceptive methods for subjects include:

   * Barrier methods, such as condom, sponge or diaphragm, combined with spermicide in foam, gel or cream;
   * Hormonal contraception (oral, intramuscular, implant or transdermal which includes Depo-Provera, Evra and Nuvaring);
   * Intrauterine device (IUD)
6. Mentally and legally capable of giving informed consent prior to any study related procedures

Exclusion Criteria:

1. Presence of systemic or localized diseases, conditions, or medications that could interfere with assessment of safety and efficacy or that compromise immune function including psoriasis
2. Subject has been diagnosed with diabetes mellitus
3. Subject has a history of keloid formation
4. Injectable common wart(s) located in areas with existing dermatologic conditions (such as psoriasis) or with an underlying inflammatory conditions (such as arthritic joints), or tattoos or implants/piercing/hardware or marking that may conceal responses or reactions are excluded from injection
5. Existing/planned pregnancy, childbirth in the past six months prior to the Baseline Visit, or breast feeding, or plan on donating eggs or sperm during the study and in the month following the last injection
6. Treatment of warts with liquid nitrogen, carbon dioxide, electrodessication, laser, surgery, simple occlusion (e.g. duct tape) salicylic or related acids, OTC treatments, cantharidin, or other treatments within 4 weeks of the Baseline Visit
7. Treatment with immunotherapy (DPCP, DNCB or other), imiquimod, 5-fluorouracil, bleomycin, podophyllin or any other wart immunotherapy or treatment designed to stimulate immune response (except for treatments already listed in exclusion criterion 6) within 12 weeks of the Baseline Visit
8. Recalcitrant warts defined as those not successfully treated by 5 or more treatments (excluding OTC treatments)
9. Abnormal (low < 5 mm or high >25 mm) baseline result to the Delayed Type Hypersensitivity (DTH) test
10. Subject has a condition or treatment resulting in being immunocompromised
11. Systemic treatment (such as oral or injected) with cimetidine, zinc supplements at a dose higher than 20 mg of elemental zinc daily or an immunosuppressive drug (such as: azathioprine, 6-mercaptopurine, methotrexate, infliximab, adalimumab, etanercept, systemic steroids, etc.) within 12 weeks of the Baseline Visit
12. Subject has used any investigational agent within 30 days prior to the Baseline Visit or within 5 half-lives of that investigational agent prior to the Baseline Visit (whichever is longer)
13. Previous treatment of warts with any type of intralesional injection with candida extract (including CANDIN)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Carpenter, DVM, PhD, Study Director — Nielsen BioSciences, Inc.
Locations (15):
- United States (15):
  - Johnson Dermatology, Fort Smith, Arkansas
  - Northwest Arkansas Clinical Trials Center PLLC, Rogers, Arkansas
  - California Dermatology and Clinical Research Institute, Encinitas, California
  - Silverberg MD Inc., Newport Beach, California
  - Metro Boston Clinical Partners, LLC, Needham, Massachusetts
  - BayState Clinical Trials, Watertown, Massachusetts
  - Hamzavi Dermatology Clinical Trials, Fort Gratiot, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Dermatology Consulting Services, High Point, North Carolina
  - Oregon Medical Research Center, Portland, Oregon
  - Austin Institute for Clinical Research Inc., Austin, Texas
  - DermResearch Inc., Austin, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - The Education and Research Foundation, Inc., Lynchburg, Virginia

REFERENCES:
- [Result] Kim KH, Horn TD, Pharis J, Kincannon J, Jones R, O'Bryan K, Myers J, Nakagawa M. Phase 1 clinical trial of intralesional injection of Candida antigen for the treatment of warts. Arch Dermatol. 2010 Dec;146(12):1431-3. doi: 10.1001/archdermatol.2010.350. No abstract available. PMID 21173332
- [Derived] Smith SR, Esch RE, Nielsen HS, Johnson SM. Randomized Phase IIa Trial of Purified Candida Antigen for Common Warts: Evaluating the Safety and Efficacy Across Multiple Dosing Regimens. Dermatol Ther (Heidelb). 2025 May;15(5):1135-1152. doi: 10.1007/s13555-025-01387-1. Epub 2025 Mar 29. PMID 40155509

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screen Fail Rate of 30% - 12% due to warts not meeting criteria, 12% due to DTH measurement not meeting criteria, 5% other reasons.
Period: Overall Study
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Started (Subjects Randomized) | 43 | 45 | 40 | 41
Completed Treatment | 30 | 34 | 32 | 30
Completed (Completed Treatment and both follow up visits) | 28 | 32 | 30 | 29
Not Completed | 15 | 13 | 10 | 12

BASELINE CHARACTERISTICS:
Population: mITT- modified Intent to Treat population consisted of subjects that received at least one post baseline measurement of the primary wart(s).
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 43 | 44 | 39 | 40 | 166
Age, Continuous [Mean (Full Range); unit: years] | 34.7 [18 to 65] | 35.6 [19 to 63] | 33.5 [18 to 62] | 30.2 [18 to 54] | 33.6 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 24 | 11 | 68
  Male | 27 | 27 | 15 | 29 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 4 | 6 | 19
  Not Hispanic or Latino | 39 | 39 | 35 | 34 | 147
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 0 | 4
  White | 41 | 40 | 30 | 37 | 148
  More than one race | 0 | 0 | 2 | 0 | 2
  Unknown or Not Reported | 0 | 3 | 2 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 43 | 44 | 39 | 40 | 166
Response (size of induration) to CANDIN injection during screening [Mean (Standard Deviation); unit: mm] — CANDIN is currently marketed in the US and was used as indicated in this study as a recall antigen for detecting delayed-type hypersensitivity (DTH) following intradermal injection of 0.1 mL.
  mm | 9.95 (4.116) | 12.09 (5.672) | 11.01 (4.534) | 10.30 (3.902) | 10.85 (4.661)
Body Weight [Mean (Standard Deviation); unit: kg] | 93.91 (28.165) | 90.30 (22.753) | 81.77 (18.977) | 83.27 (21.929) | 87.54 (23.629)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 30.75 (8.812) | 29.11 (6.291) | 27.85 (6.461) | 27.42 (7.486) | 28.83 (7.392)
Location of Common Warts [Number; unit: each]
  Left Hand | 29 | 21 | 25 | 35 | 110
  Right Hand | 36 | 36 | 26 | 37 | 135
  Left Arm | 6 | 4 | 1 | 5 | 16
  Right Arm | 0 | 7 | 3 | 2 | 12
  Left Leg | 3 | 1 | 3 | 5 | 12
  Right Leg | 4 | 1 | 3 | 1 | 9
  Left Foot (excluding sole) | 1 | 0 | 3 | 2 | 6
  Right Foot (excluding sole) | 3 | 0 | 1 | 2 | 6
Area of Primary Injected Wart [Mean (Full Range); unit: mm^2] | 32.19 [9.4 to 233.3] | 41.47 [7.1 to 238.8] | 36.95 [7.1 to 150.8] | 27.66 [7.1 to 92.3] | 34.68 [7.1 to 238.8]
Age of Primary Injected Wart(s) [Mean (Full Range); unit: weeks] | 228.9 [12 to 1560] | 202.0 [14 to 1040] | 174.7 [16 to 1092] | 196.8 [12 to 670] | 201.3 [12 to 1560]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Complete Resolution of a Primary Injected Wart(s) at Any Treatment or Follow-up Visit
Description: Complete resolution of a wart was defined as the absence of visible or measurable presence of the wart
Time Frame: 45 weeks
Population: Modified Intent to Treat (mITT) - subjects that received at least one post baseline measurement of the primary wart(s)
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 43 | 44 | 39 | 40
Participants | 16 | 29 | 31 | 29
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort 1; Test type: Superiority; p = 0.0329, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.5706, 95% CI 2-sided [1.0184 to 2.4223]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort 2; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.8926, 95% CI 2-sided [1.2722 to 2.8156]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort 3; Test type: Superiority; p = 0.0052, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.7319, 95% CI 2-sided [1.1602 to 2.5854]

2. Secondary Outcome: Number of Subjects With a Complete Resolution of All Common Warts at Any Treatment or Follow-up Visit
Description: Complete resolution of a wart was defined as the absence of visible or measurable presence of the wart
Time Frame: 45 weeks
Population: mITT - Subjects that received at least one post baseline measurement of the primary wart(s)
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 43 | 44 | 39 | 40
Participants | 7 | 12 | 20 | 12
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort 1; Test type: Superiority; p = 0.4307, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.3828, 95% CI 2-sided [0.6191 to 3.0883]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort 2; Test type: Superiority; p = 0.0014, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 2.8908, 95% CI 2-sided [1.4169 to 5.8978]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort 3; Test type: Superiority; p = 0.0451, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 3.0000, 95% CI 2-sided [0.9281 to 9.6975]

3. Secondary Outcome: Number of Subjects With Complete Resolution of Primary Injected Wart(s) at the 4 Month Follow-up Visit
Description: Complete resolution of a wart was defined as the absence of visible or measurable presence of the wart
Time Frame: 4 month follow up visit at 45 weeks
Population: mITT - Subjects that received at least one post baseline measurement of the primary wart(s)
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 43 | 44 | 39 | 40
Participants | 16 | 20 | 27 | 20

4. Secondary Outcome: Number of Injection Visits Needed to Obtain Complete Resolution of the Primary Injected Wart(s)
Description: Complete resolution of a wart was defined as the absence of visible or measurable presence of the wart
Time Frame: 45 weeks
Population: mITT. Subjects that received at least one post baseline measurement of the primary wart(s). Cohort 3 values represent resolution of largest primary wart
Measure: Median (95% Confidence Interval); unit: injection visits
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 43 | 44 | 39 | 40
injection visits | 10 [10 to 10] | 5 [3 to 10] | 5 [3 to 10] | 4 [3 to 8]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort 1; Test type: Superiority; p = 0.0027, Regression, Cox; Cox Proportional Hazard = 2.7553, 95% CI 2-sided [1.4211 to 5.3419]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort 2; Test type: Superiority; p = 0.0008, Regression, Cox; Cox Proportional Hazard = 3.1516, 95% CI 2-sided [1.6148 to 6.1509]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort 3; Test type: Superiority; p = 0.0003, Regression, Cox; Cox Proportional Hazard = 3.3257, 95% CI 2-sided [1.7263 to 6.4070]

5. Secondary Outcome: Number of Injection Visits for >50% Reduction in Area of the Primary Injected Wart(s)
Time Frame: 45 weeks
Population: mITT - Subjects that received at least one post baseline measurement of the primary wart(s)
Measure: Median (95% Confidence Interval); unit: injection visits
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 43 | 44 | 39 | 40
injection visits | 9.0 [6.0 to 10.0] | 3.0 [2.0 to 4.0] | 2.0 [2.0 to 4.0] | 2.0 [1.0 to 2.0]

6. Secondary Outcome: Number of Injection Visits to >50% Reduction in the Total Area of All Measured Warts
Time Frame: 45 weeks
Population: mITT - Subjects that received at least on post baseline measurement of the primary wart(s)
Measure: Median (95% Confidence Interval); unit: injection visits
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 43 | 44 | 39 | 40
injection visits | 10.0 [8.0 to NA] — Value cannot be estimated due to insufficient number of participants with events | 5.0 [4.0 to 9.0] | 4.0 [2.0 to 6.0] | 3.0 [2.0 to 4.0]

7. Secondary Outcome: Number of Subjects With Scarring at the Site of Resolved Primary and Non-primary Injected Wart(s)
Description: Scarring at any visit, many reports were transient being noted at only one or two visits and noted as resolving during the course of the study
Time Frame: 45 weeks
Population: mITT - Subjects that received at least one post baseline measurement of the primary wart(s)
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 18 | 28 | 31 | 33
Participants | 1 | 7 | 3 | 3

8. Secondary Outcome: Number of Subjects With Hypopigmentation at the Site of Resolved Primary and Non-primary Injected Wart(s)
Time Frame: 45 weeks
Population: Only mITT subjects with complete resolution of warts included in this endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 18 | 28 | 31 | 33
Participants | 0 | 1 | 1 | 2

9. Secondary Outcome: Number of Subjects With Injection Site Reactions With Frequency Greater Than 5%
Time Frame: 45 weeks
Population: Safety Population- All randomized subjects who received at least one intralesional dose of study medication. Subjects experiencing multiple types of reactions were counted once for each type, but only once across all reactions.
Measure: Number; unit: participants
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 43 | 45 | 40 | 41
participants
  Tenderness | 27 | 42 | 40 | 39
  Pain | 15 | 41 | 35 | 39
  Pruritis/Itching | 13 | 36 | 32 | 33
  Edema/Swelling | 9 | 17 | 27 | 23
  Erythema/Redness | 3 | 18 | 25 | 23
  Peeling | 1 | 3 | 2 | 8
  Scarring | 1 | 6 | 2 | 2

10. Other Pre Specified Outcome: Association Between the Age of the Largest Primary Injected Wart and Complete Resolution of the Largest Primary Injected Wart
Description: Complete resolution of a wart was defined as the absence of visible or measurable presence of the wart
Time Frame: 45 weeks
Population: mITT- Subjects that received at least one post baseline measurement of the primary wart(s)
Measure: Number; unit: number of warts resolved
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 43 | 44 | 39 | 40
number of warts resolved | 18 | 29 | 31 | 29
Statistical Analysis 1: Comparison: Pooled Placebo; Using a logistic regression model for complete resolution status of largest primary injected wart (yes vs no) with wart age as a covariate; Test type: Superiority; p = 0.4824, Regression, Logistic; Odds Ratio (OR) = 0.999, 95% CI 2-sided [0.997 to 1.001] — An odds ratio < 1 indicates that the age of the wart is negatively correlated with positive treatment outcome and vice versa
Statistical Analysis 2: Comparison: Cohort 1; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.5007, Regression, Logistic; Odds Ratio (OR) = 1.001, 95% CI 2-sided [0.998 to 1.004] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Cohort 2; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.0219, Regression, Logistic; Odds Ratio (OR) = 0.993, 95% CI 2-sided [0.987 to 0.999] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: Cohort 3; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.8267, Regression, Logistic; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.995 to 1.004] — [estimate comment as in outcome 10, analysis 1]

11. Other Pre Specified Outcome: Association Between the Age of the Primary Injected Wart and the Recurrence of Any Resolved Wart at Any Visit.
Time Frame: 45 weeks
Population: mITT - subjects that received at least one post baseline measurement of the primary wart(s)
Measure: Number; unit: wart recurrences
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 20 | 33 | 34 | 34
wart recurrences | 5 | 14 | 13 | 24
Statistical Analysis 1: Comparison: Pooled Placebo; Using a logistic regression model for recurrence status of any resolved wart (yes vs no) with age of the largest primary injected wart as a covariate; Test type: Superiority; p = 0.1657, Regression, Logistic; Odds Ratio (OR) = 0.964, 95% CI 2-sided [0.915 to 1.015] — An odds ratio > 1 indicates that the age of the largest primary injected wart is positively correlated with the recurrence of any resolved wart and vice versa
Statistical Analysis 2: Comparison: Cohort 1; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.8168, Regression, Logistic; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.997 to 1.003] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Cohort 2; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.4183, Regression, Logistic; Odds Ratio (OR) = 0.998, 95% CI 2-sided [0.993 to 1.003] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Cohort 3; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.5572, Regression, Logistic; Odds Ratio (OR) = 1.001, 95% CI 2-sided [0.997 to 1.006] — [estimate comment as in outcome 11, analysis 1]

12. Other Pre Specified Outcome: Summary of Complete Resolution of the Largest Primary Wart and Type of Treatment History
Description: Complete resolution of a wart was defined as the absence of visible or measurable presence of the wart
Time Frame: 45 weeks
Population: mITT- Subjects that received at least one post baseline measurement of the primary wart(s). A subject may belong to more than one prior treatment types. As defined in the Statistical Analysis Plan, Cohorts 1 and 3 were combined for this exploratory endpoint (0.3 mL injected into each wart)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 and Cohort 3: 0.3 mL of CANDIN administered intralesionally in the largest common wart (Cohort 1) and multiple common warts (Cohort 3)
  CANDIN: Candida albicans Skin Test Antigen for Cellular Hypersensitivity
Arm/Group | Pooled Placebo | Cohort 1 and Cohort 3 | Cohort 2
Number analyzed (Participants) | 43 | 84 | 39
Participants
  Naive | 12 | 24 | 11
  Cryotherapy | 6 | 27 | 17
  Surgery | 0 | 1 | 0
  Salicylic acid | 1 | 12 | 6
  Other | 0 | 1 | 3

13. Other Pre Specified Outcome: The Effect of the Treatment History on the Number of Recurrences of Resolved Primary Warts
Time Frame: 45 weeks
Population: mITT - Subjects that received at least one post baseline measurement of the primary wart(s). A subject may belong to more than one prior treatment types. As defined in the Statistical Analysis Plan, Cohorts 1 and 3 were combined for this exploratory endpoint (0.3 mL injected into each wart)
Measure: Number; unit: Number of warts
Arm/Group | Pooled Placebo | Cohort 1 and Cohort 3 | Cohort 2
Number analyzed (Participants) | 2 | 26 | 7
Number of warts
  Naive | 2 | 11 | 3
  Cryotherapy | 0 | 13 | 4
  Surgery | 0 | 0 | 0
  Salicylic Acid | 0 | 7 | 2
  Other | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Events during or after the first wart injection through the last visit, up to 45 weeks
Description: Incidence of Treatment Emergent, Non-Injection Site Reactions
Arm/Group | Pooled Placebo | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/45 | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/45 | 2/40 | 1/41
Other Adverse Events (participants affected / at risk) | 32/43 | 33/45 | 34/40 | 33/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=43) | Cohort 1 (N=45) | Cohort 2 (N=40) | Cohort 3 (N=41)
Pancreatitis, Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Brain Abcess (Infections and infestations) | 0 | 0 | 1 (1) | 0
Mediastinal Abcess (Infections and infestations) | 0 | 0 | 1 (1) | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=43) | Cohort 1 (N=45) | Cohort 2 (N=40) | Cohort 3 (N=41)
Headache (Nervous system disorders) | 16 | 15 | 15 | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 14 | 14 | 13
Fatigue (General disorders) | 15 | 12 | 14 | 13
Diarrhoea (Gastrointestinal disorders) | 7 | 13 | 9 | 9
Nausea (Gastrointestinal disorders) | 3 | 6 | 9 | 11
Influenza (Infections and infestations) | 9 | 4 | 6 | 13
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2 | 6 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 6
Influenza Like Illness (General disorders) | 2 | 5 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 3
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 4
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3 | 1
Pyrexia (General disorders) | 3 | 0 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 2 | 1
Migraine (Nervous system disorders) | 0 | 1 | 2 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT02393417/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT02393417/SAP_001.pdf